CLINICAL TRIAL: NCT03146364
Title: Evaluation of Executive Function With Static and Dynamic Shopping Assignment in Virtual Reality Among People With Schizophrenia
Brief Title: Evaluation of Executive Function With Virtual Reality Among People With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Alon Reshef, Head of psychiatry, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HaEmekAlon
Record Dates: First submitted 2017-04-01; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: Virtual Reality
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospitalization patients (Experimental): patients in psychiatric hospitalization will take part in tests at Virtual Reality - Virtual Interactive Supermarket environment (diagnosis)
  Interventions: Device: Virtual Reality - Virtual Interactive Supermarket
- Ambulatory patients (Experimental): patients being treated in a clinic will take part in tests at Virtual Reality - Virtual Interactive Supermarket environment (diagnosis)
  Interventions: Device: Virtual Reality - Virtual Interactive Supermarket

INTERVENTIONS:
Device: Virtual Reality - Virtual Interactive Supermarket — SeeMe is a PC based, innovative, comprehensive, clinician-controlled exercise and diagnostic system. SeeMe is designed to aid the rehabilitation process, and track patients' progress.
  Virtual Interactive Supermarket- one of the SeeMe Tasks, the user need to buy products by according to specific instruction
  Other Names: SeeMe

SUMMARY:
This Cross-sectional Study Included Patients that diagnosed with schizophrenia, aged 18-55, 20 of which hospitalized in mental health department and 20 in medical follow-up.

Different test will be administered, in two or three sessions, to evaluate cognitive ability, function ability and participation.

The results of the VIS shopping task performance (statically & dynamically) and its correlation with the cognitive and function tests as well as the participation questionnaire will be examined. These findings will indicate whether the shopping task is valid to assess executive functions for people with schizophrenia and whether it is ecologically valid.

DETAILED DESCRIPTION:
Background:

Schizophrenia often reflect by decrease in executive functions that may cause difficulty in Instrumental Activities of Daily Living (IADL). We've found it very difficult to simulate these functions with the existing tools in the clinic and to assess IADL accordingly.

The use of Virtual Reality (VR) became popular in the last decade to overcome these limitations in clinical practice and assessment of functioning in IADL. VR is a computer program that simulates a functional environment in which the subject impacts on events through various actions. Recent studies indicated that VR can be used to assess cognitive abilities and functioning of population with schizophrenia. As far as we know, no researches were performed using Virtual Interactive Shopping (VIS) in this population, nor did dynamic evaluation was used to identify potential learning abilities. The aim of this study is to examine the validity of the shopping task in the VIS, performed statically and dynamically, in order to assess executive function, and the ability to reflect cognitive, functional and participation ability among people that diagnosed with schizophrenia.

Method:

This Cross-sectional Study Included Patients that diagnosed with schizophrenia, aged 18-55, 20 of which hospitalized in mental health department and 20 in medical follow-up.

Different test will be administered, in two or three sessions, to evaluate cognitive ability, function ability and participation.

The results of the VIS shopping task performance (statically & dynamically) and its correlation with the cognitive and function tests as well as the participation questionnaire will be examined. These findings will indicate whether the shopping task is valid to assess executive functions for people with schizophrenia and whether it is ecologically valid.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or Scizoeffective diagnosis, Hebrew language proficiency, three weeks of anti-psychotic drug treatment

Exclusion Criteria:

* score of under 70 in the 3MS (screen test), physical disability, neurological diagnosis (ex. dementia)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Modified 4 item test | through study completion, an average of 1 year
  "buy" 4 items with budget constraints, using the VIS

SECONDARY OUTCOMES:
Revised Observed Tasks of Daily Living (OTDL-R) | through study completion, an average of 1 year
  evaluation of IADL using various tasks include problem solving
Executive Function Performance Test (EFPT) | through study completion, an average of 1 year
  executive function assessment using 5 different tasks
Trail Making Test A & B (TMT) | through study completion, an average of 1 year
  The Trail Making Test is an accessible neuropsychological instrument that provides the examiner with information on a wide range of cognitive skills and can be completed in 5-10 min.
The positive and negative syndrome scale (PANSS) | through study completion, an average of 1 year
  The Positive and Negative Syndrome Scale (PANSS) was developed out of the need for a well-operationalized method of assessing these syndromes in schizophrenia, including their relationship to one another and to global psychopathology
Adults Subjective Assessment of Participation | through study completion, an average of 1 year
  participation questionnaire that examine the level of engagement in different occupations

IPD SHARING:
Plan to Share IPD: No